CLINICAL TRIAL: NCT04059952
Title: Mechanism of Action of Electroconvulsive Therapy
Acronym: MoA-ECT
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joan A Camprodon, MD MPH PhD, Chief of Division of Neuropsychiatry, Director of TMS Clinic, Director of Lab for Neuropsychiatry and Neuromodulation, Massachusetts General Hospital
Other Study IDs: 2012P001430
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Unipolar Depression; Bipolar Depression
Keywords: Electroconvulsive Therapy; Magnetic Resonance Imaging
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Unipolar Depression: Patients diagnosed with Major Depressive Disorder.
  Interventions: Device: Electroconvulsive Therapy
- Bipolar Depression: Patients diagnosed with Bipolar I or II.
  Interventions: Device: Electroconvulsive Therapy
- Healthy Control: Patients without psychiatric diagnoses.

INTERVENTIONS:
Device: Electroconvulsive Therapy — Electrical currents are passed through the brain to intentionally trigger a controlled seizure in order to produce a therapeutic change in neuro-chemistry and circuitry.
  Groups: Bipolar Depression; Unipolar Depression

SUMMARY:
This is an observational neuroimaging study assessing the effects of ECT on the brains of patients with unipolar and bipolar depression.

DETAILED DESCRIPTION:
This project aims to use functional connectivity magnetic resonance imaging (fcMRI) to study patients with unipolar and bipolar depression receiving ECT. Patients will be scanned before and after a full course of ECT and clinical measures for depression severity and memory will be obtained at the same times.The project has the following aims and hypothesis: (1) to determine the therapeutic antidepressant mechanism of action of ECT at the circuit level (2) to determine the mechanism of action of iatrogenic amnesia caused by ECT at the circuit level (3) to study the use of fcMRI as a state biomarker for depression (4) to study the use of fcMRI as a predictor of response for depression.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females Between Ages of 18 and 65
* Diagnosis of Major Depressive Disorder without Psychotic Features or Bipolar I/II
* Requiring ECT Treatment as Part of Psychiatric Care

Exclusion Criteria:

* Comorbid diagnoses of Major Depressive Disorder with Psychotic Features, Schizoaffective Disorder, Schizophrenia or Dementia
* History of Psychosis
* Substance Use Disorder (Abuse or Dependence) with Active Use Within Last 6 Months
* Severe or Unstable Medical Illness
* Medical Contraindication to Anesthesia or ECT (e.g., Recent Myocardial Infarction)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and Female Patients with Unipolar or Bipolar Depression Between the Ages of 18 and 65 Being Treated with ECT as Part of Outpatient Psychiatric Care, or Healthy Controls.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in Functional Connectivity of Key Nodes | Through Treatment Completion, Average of 2 Months
  Measured by Magnetic Resonance Imaging, Key Nodes include Subgenual Cingulate, Dorsal Anterior Cingulate, Nucleus Accumbens, Hippocampus, Amygdala and Dorsolateral Prefrontal Cortex

SECONDARY OUTCOMES:
Changes in Functional Connectivity of Memory Circuits | Through Treatment Completion, Average of 2 Months
  Measured by Magnetic Resonance Imaging, Memory Circuits Include Hippocampus and Dorsolateral Prefrontal Memory Hubs

CONTACTS AND LOCATIONS:
Overall Officials: Joan Camprodon, MD MPH PHD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All identifying information (e.g., name, medical record number, date of birth) will be removed from data that will be shared with other researchers or research databases. It will not be possible to link the information back to the participant.
Time Frame: Data will become available at study completion for an undefined amount of time.
Access Criteria: Data will be accessible by researchers who have access to research databases at the NIH.